CLINICAL TRIAL: NCT06602050
Title: Determination of the Relationship Between Maximum Inspiratory Pressure, Grip Strength and Physical Functional Status in Mechanically Ventilated Patients
Brief Title: Maximum Inspiratory Pressure, Grip Strength and Physical Functional Status Relationship in MV Patients
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: SB Goztepe Prof Suleyman Yalcin City Hospital (Unknown)
Responsible Party: Principal Investigator, Mehmet Burak Uyaroğlu, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: sagbilimuni
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Mechanical Ventilation Complication; Intensive Care Medicine
Keywords: Mechanical Ventilation; Maximal Inspiratory Pressure; handgrip strength; Physical function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HG and NIF: The cohort will consist of cooperative mechanically ventilated (MV) patients. In this patient group, the relationships between negative inspiratory force (NIF), handgrip strength (HG), and physical functional status will be examined.
  Interventions: Other: HG and NIF

INTERVENTIONS:
Other: HG and NIF — In mechanically ventilated patients, handgrip strength, the Negative Inspiratory Force (NIF) value obtained via the ventilator, and physical function through various tests will be assessed.

SUMMARY:
The maximal inspiratory pressure or negative inspiratory force values is a parameter that measures the functional ability of the respiratory system. The ability to reduce the risk of atelectasis, effective coughing and mobilization of airway secretions is directly proportional to the magnitude of this value. Grip strength is a parameter that noninvasively assesses functional status in critical care patients.Respiratory muscles work in a complex interaction with peripheral muscles. This dynamic relationship has been described in many populations.The aim of this study was to determine the relationship between maximum inspiratory pressure and grip strength and physical functional status in mechanical ventilator patients.

DETAILED DESCRIPTION:
Progressive inadequate ventilation results in multiple organ dysfunction due to impaired oxygenation and subsequent hypoxia. Additionally, the combined effects of reduced exercise capacity and increased oxidative stress contribute to cardiovascular failure, further immobilization, increased peripheral muscle weakness, and a diminished quality of life. From this standpoint, there is a dynamic interaction between the respiratory muscles and peripheral striated muscles; strengthening one muscle group positively influences the other. Respiratory muscle strength is closely related to both limb muscle strength and endurance. Therefore, it is essential to assess not only respiratory but also peripheral muscle strength in mechanically ventilated patients.

Maximum Inspiratory Pressure (MIP) and Maximum Expiratory Pressure (MEP) are functional units used to assess respiratory muscle strength. In this context, various measurement methods developed to determine MIP and MEP provide valuable insights into the condition of patients' respiratory muscles. Although invasive methods are sometimes used to evaluate respiratory muscle strength in mechanically ventilated patients, simple bedside measurements are often sufficient. One such method, particularly for ventilator-dependent patients, utilizes the negative inspiratory pressure value available through the ventilator's software features. In this procedure, the intensive care unit clinician instructs the patient to perform a strong inspiratory effort against a "closed circuit" within the system, and the resulting pressure serves as an indicator of inspiratory muscle strength. It is crucial that the patient is informed about the absence of airflow during this procedure and that they are cooperative.

Peripheral muscle strength is typically assessed using muscle strength tests or isokinetic evaluations. Additionally, grip strength measurement serves as a non-invasive indicator of both functional status and peripheral muscle strength in patients on mechanical ventilation .Respiratory muscles work in a complex interaction with peripheral muscles.This dynamic relationship has been described in many populations. In certain disease groups, peripheral muscle strength has been assessed through grip strength, while respiratory muscle strength was measured using maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) values, allowing for the determination of the relationship between these two muscle groups. Typically, MIP is measured in the literature using manometers and specialized devices. However, this study was designed to measure MIP using the negative inspiratory pressure value-equivalent to maximal inspiratory pressure-directly from the mechanical ventilation device, without the use of external equipment and without disconnecting the patient from the respiratory circuit.The aim of this study is to determine the relationship between maximal inspiratory pressure, grip strength, and physical functional status in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable
* Consciousness level sufficient to follow commands
* Patients with functionally intact extremities

Exclusion Criteria:

* Patients with neurological disorders (central or peripheral)
* Patients with craniocerebral injury
* Patients using medications that affect muscle tone
* Patients using sedative agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Conscious and cooperative patients receiving mechanical ventilation (MV) support
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
Assessment of Inspiratory Pressure | At baseline, on the day of enrollment
  Negative Inspiratory Force (NIF), also known as Maximal Inspiratory Pressure (MIP), is an indicator of respiratory muscle strength. To measure Negative Inspiratory Pressure, the expiratory hold button on the device will be pressed for 20 seconds. After this procedure, the patient will be instructed to take deep breaths voluntarily. In the resulting graph, the y-axis will display airway pressure (Paw). The most negative value on the y-axis, when added to the Positive End-Expiratory Pressure (PEEP) value, will determine and record the individuals maximal inspiratory value.
Assessment of physical function | At baseline, on the day of enrollment
  The PFIT (Physical Function ICU Test) evaluates four key physical function components, each reported as a separate outcome measure. These components include standing ability, the level of assistance required for sit-to-stand, knee extension strength (assessed bilaterally), and the number of steps taken in one minute. MRC (Medical Research Council) muscle strength scale is used to determine knee flexion, elbow flexion and shoulder abduction muscle strength. Each parameter is scored between 0 and 3. A total score of 12 indicates that the person moves without support. These separate measures provide a comprehensive assessment of a patient's physical capacity in the ICU.Each parameter is scored between 0 and 3. A total score of 12 indicates that the person moves without support.
Assesment of Hand Grip Measurement | At baseline, on the day of enrollment
  Handgrip strength will be measured in pounds (lbs) using the Jamar Hydraulic Hand Dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Aytekin, ICU Consultant, Study Chair — Goztepe Prof Dr Suleyman Yalcın City Hospital; Esra Pehlivan, Ass. Prof., Study Director — Saglik Bilimleri Universitesi; Mehmet Burak Uyaroglu, PhD(c). PT, Principal Investigator — Saglik Bilimleri Universitesi; Nezihe Ciftaslan Goksenoglu, ICU Consultant, Study Chair — Goztepe Prof Dr Suleyman Yalcın City Hospital
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)